CLINICAL TRIAL: NCT00715117
Title: The Efficacy of Low Dose Naltrexone Therapy in Children With Crohn's Disease
Acronym: LDN-Ped
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PSU-IRB-27793
Record Dates: First submitted 2008-07-14; First posted 2008-07-15 (Estimated); Results first posted 2013-05-30 (Estimated); Last update posted 2018-09-06 (Actual); Status verified 2013-05

CONDITIONS: Crohn's Disease
Keywords: children; pediatric; Crohn's Disease; naltrexone; LDN; IBD; Inflammatory bowel disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Naltrexone; vivitrol; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sugar pill (Placebo Comparator): Subjects will receive placebo for for the first 8 weeks administered orally one time daily. After 8 weeks placebo treated subjects are then crossed over to active drug naltrexone 0.1 mg/kg not to exceed 4.5 mg PO once daily for an additional 8 weeks.
  Interventions: Other: Placebo, sugar pill
- Naltrexone (Experimental): Naltrexone 0.1 mg/kg (not to exceed 4.5mg) once a day orally either in capsules or liquid blinded for 8 weeks followed by open-labeled naltrexone for an additional 8 weeks. Safety and toxicity will be compared to placebo. Also change in Crohn's activity index scores of naltrexone to placebo are compared.
  Interventions: Drug: Naltrexone

INTERVENTIONS:
Drug: Naltrexone — Naltrexone 0.1 mg/kg (not to exceed 4.5mg) once a day orally for 16 weeks
  Other Names: Revia, Vivitrol
  Arms: Naltrexone
Other: Placebo, sugar pill — Placebo -Sugar pill or liquid identical to active drug in appearance and taste given by mouth at bedtime once daily
  Other Names: sugar pill
  Arms: Sugar pill

SUMMARY:
It is hypothesized that oral naltrexone will improve inflammation of the bowel by increasing endogenous enkephalin levels in subjects with active Crohn's disease. This is especially important in children who often are suffering from nutritional deprivation which retards their growth.

The key objectives are to:

1. Evaluate the effects of low dose naltrexone in children with Crohn's Disease by using the Pediatric Crohn's Disease Activity Index (PCDAI), plasma inflammatory markers, weight, and pediatric quality of life survey.
2. To determine the safety and toxicity of low dose naltrexone in pediatric subjects with active Crohn's Disease.
3. Assess the potential mechanism by which naltrexone exerts its action by measuring plasma opioid (enkephalin and endorphin levels) and proinflammatory cytokines.

DETAILED DESCRIPTION:
The present proposal is designed as double-blinded placebo controlled study involving 30 children between 6-17 years of age with active Crohn's disease. Children will be treated with either naltrexone or placebo for the first 8 weeks then all subjects will receive active naltrexone drug the last 8 weeks. A one month follow-up appointment will be scheduled 4-weeks after completion of the active drug for safety and to assess Crohn's activity. Low dose naltrexone (LDN) will be dispensed in either capsules at a dose of 4.5 mg for those ages 10 years or older and in liquid form at 0.1 mg/kg for those under age of 10 or less than 45 kg. Half of the subjects in the first 8 weeks will be randomized to placebo which will be either capsules filled with avicel (see section 6.0) or diluent (flavored water) if in liquid form. Children are eligible who are not of child-bearing potential or are using two means of effective birth control, have a Pediatric Crohn's Disease Activity Index (PCDAI) of at least 31 points, and have the confirmed diagnosis of Crohn's disease by either endoscopic or radiographic tests.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must give written informed consent by parent or guardian
* Male or female subjects, > 6 - 17 years
* Patients must have endoscopic or radiographic confirmed Crohn's Disease.
* Patients must have a Pediatric Crohn's Disease Activity Index (PCDAI) of at least 31.

Exclusion Criteria:

* Adolescent women of childbearing potential and / or sexually active unless surgically sterile or using adequate contraception (either IUD, oral or deport contraceptive, or barrier plus spermicide), and willing and able to continue contraception for 3 months after the completion of the study.
* Adolescent women who are pregnant or breastfeeding
* Subjects with an ostomy or ileocolic anastomosis from surgery as these operations interfere with the PCDAI assessment
* Subjects taking tacrolimus, cyclosporin, mycophenolate, or anti-TNF-α therapy must be discontinued 4 weeks prior to study initiation.
* Patients with abnormal liver function tests
* Prednisone greater than 10 mg or > 0.2 mg/kg orally

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jill P Smith, MD, Principal Investigator — Pennsylvania State University College of Medicine
Locations (1):
- Penn State University hershey Medical center, Hershey, Pennsylvania, United States

REFERENCES:
- [Background] Smith JP, Stock H, Bingaman S, Mauger D, Rogosnitzky M, Zagon IS. Low-dose naltrexone therapy improves active Crohn's disease. Am J Gastroenterol. 2007 Apr;102(4):820-8. doi: 10.1111/j.1572-0241.2007.01045.x. Epub 2007 Jan 11. PMID 17222320
- [Background] Smith JP, Bingaman SI, Ruggiero F, Mauger DT, Mukherjee A, McGovern CO, Zagon IS. Therapy with the opioid antagonist naltrexone promotes mucosal healing in active Crohn's disease: a randomized placebo-controlled trial. Dig Dis Sci. 2011 Jul;56(7):2088-97. doi: 10.1007/s10620-011-1653-7. Epub 2011 Mar 8. PMID 21380937
- [Result] Smith JP, Field D, Bingaman SI, Evans R, Mauger DT. Safety and tolerability of low-dose naltrexone therapy in children with moderate to severe Crohn's disease: a pilot study. J Clin Gastroenterol. 2013 Apr;47(4):339-45. doi: 10.1097/MCG.0b013e3182702f2b. PMID 23188075
- See also: Penn State College of Medicine- Clinical Trials Office Site — http://www.hmc.psu.edu/clinicaltrials/studies/gi/index.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 14 subjects were enrolled in this pilot trial and 2 were screen failures and not randomized or treated
Pre-assignment Details: The 2 subjects who were screen failures had PCDAI scores less than 30.
Groups:
- A: Placebo Then Naltrexone: Subjects will receive placebo for for the first 8weeks then be crossed over to active drug naltrexone for the last 8 weeks
- B: Naltrexone Then Naltrexone: Naltrexone 0.1 mg/kg (not to exceed 4.5mg) once a day for 8 weeks followed by the same treatment for an additional 8 weeks
Period: Overall Study
Arm/Group | A: Placebo Then Naltrexone | B: Naltrexone Then Naltrexone
Started | 6 | 6
Completion fo 8 Week Study | 6 | 6
Completed | 6 | 5 (One subject flared and was rescued with steroids)
Not Completed | 0 | 1
Not completed — Crohn's flare and rescue with steroids | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- A: Placebo Control Group: Subjects will receive placebo for for the first 8weeks then be crossed over to active drug for the last 8 weeks
- B: Naltrexone, Active Drug Group: Naltrexone 0.1 mg/kg (not to exceed 4.5mg) once a day for 16 weeks
- Total: Total of all reporting groups
Arm/Group | A: Placebo Control Group | B: Naltrexone, Active Drug Group | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6 | 6 | 12
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 12.2 (3.31) | 13 (3.22) | 12.5 (3.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 1 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 12
Pediatric Crohn's Disease Activity Index (PCDAI) score [Mean (Full Range); unit: score] — The PCDAI score is a number unit that is calculated from symptoms scores by the subject over a 7-day period prior to the visit, laboratory values, height & weight, and physical exam findings. A score of 10 and under denotes "remission". Mild disease (score of 11-30); moderate disease (score of 31-45), a severe disease (scores greater than 45. A decline of 10 points or more is considered "response to therapy". The score can range from 0 to >60 Patient must have a PCDAI score of equal or greater than 30 to qualify for this study (i.e., moderate to severe disease).
  score | 45 [35 to 52.5] | 38.3 [30 to 57] | 41.7 [30 to 57]

OUTCOME MEASURES:

1. Secondary Outcome: Pediatric Crohn's Disease Activity Index Score (PCDAI)
Description: Secondary outcome was efficacy on clinical activity. Mean pretreatment PCDAI scores in patients had moderate to severe disease activity at baseline were compared between those who received placebo for 8 weeks and those who received active experimental drug, naltrexone.
  The PCDAI score is a number unit that is calculated from symptoms scores by the subject over a 7-day period prior to the visit, laboratory values, height & weight, and physical exam findings. A score of 10 and under denotes "remission". Mild disease (score of 11-30); moderate disease (score of 31-45), a severe disease (scores greater than 45. A decline of 10 points or more is considered "response to therapy". The score can range from 0 to >60 Patient must have a PCDAI score of equal or greater than 30 to qualify for this study (i.e., moderate to severe disease).
Time Frame: Pretreatment and 8 weeks
Population: The power calculations were performed using STPLAN version 4.1. The current investigation was designed as a pseudo-cross over study to increase the number of participants. In the proposed study, it was assumed that 80% would respond to naltrexone and that no more than 25% of the placebo.
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- All Participants Pretreament: All participants prior to receiving placebo or naltrexone at week 0
- Placebo: Patients were treated with a placebo (sugar pill)for 8 weeks.
- Naltrexone: Includes all Naltrexone treated participants 8 weeks of treatment.
Arm/Group | All Participants Pretreament | Placebo | Naltrexone
Number analyzed (Participants) | 12 | 6 | 12
units on a scale | 34.2 (3.3) | 30 (4.9) | 21.7 (3.9)
Statistical Analysis 1: Comparison: All Participants Pretreament vs Naltrexone; Test type: Superiority or Other; p = 0.005, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Naltrexone; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

2. Secondary Outcome: Change in Quality of Life Scores From Baseline to After 8 Weeks of Naltrexone Therapy
Description: IMPACT III was a pediatric Crohn's specific quality of life survey used in this study. It examines five major categories influencing the quality of life in children with Crohn's disease including bowel symptoms, systemic symptoms, emotional well-being, social well-being, and body image perception. The IMPACT-III uses 5-point Likert scale ranging from 1 to 5 for all answers. The outcome score ranges from 35 to 175, with higher scores suggesting better quality of life. So an increase in score denotes improved Quality of life.
Time Frame: 16 weeks
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- Baseline: Quality of life values in all subjects at baseline before receiving placebo or naltrexone.
- Week 16: Quality of life survey values in all subjects determined at week 16 after all 12 participants had received naltrexone for either 8 or 16 weeks.
Arm/Group | Baseline | Week 16
Number analyzed (Participants) | 12 | 12
units on a scale
  Bowel symptoms | 20 (2.1) | 23 (1.9)
  Social well-being | 40 (0.9) | 45 (0.8)
  Emotional Well-being | 20 (1.6) | 24 (1.5)
  Systemic symtoms | 9.8 (0.2) | 10.1 (0.2)
  Body image | 10.2 (0.2) | 10.3 (0.2)
Statistical Analysis 1: Comparison: Baseline vs Week 16; Bowel symptoms; Test type: Superiority or Other; p > 0.05, t-test, 2 sided
Statistical Analysis 2: Comparison: Baseline vs Week 16; Social well-being; Test type: Superiority or Other; p = 0.035, t-test, 2 sided
Statistical Analysis 3: Comparison: Baseline vs Week 16; Emotional well-being; Test type: Superiority or Other; p > 0.05, t-test, 2 sided
Statistical Analysis 4: Comparison: Baseline vs Week 16; Test type: Superiority or Other; p = 0.035, t-test, 2 sided — Systemic symptoms
Statistical Analysis 5: Comparison: Baseline vs Week 16; Body Image; Test type: Superiority or Other; p > 0.05, t-test, 2 sided

3. Primary Outcome: Number of Patients Reporting Side Effects
Description: Using adverse events and laboratory values Safety & toxicity were evaluated between those on placebo for 8 weeks and those on naltrexone for either 8 or 16 weeks.
Time Frame: 8 weeks or 16 weeks
Population: The Fisher Exact Test was used to evaluate the number of side effects reported between placebo and naltrexone groups. The Student T-test was used to evaluate the differences between the mena values of laboratory tests.
Measure: Number; unit: participants
Groups:
- Placebo: These subjects received placebo for 8 weeks by mouth daily.
- Naltrexone: These subjects were treated with naltrexone at a dose 0.1 mg/kg not to exceed 4.5 mg po daily for either 8 or 16 weeks.
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 6 | 12
participants
  Sleep disturbance | 2 | 2
  Unusal Dreams | 0 | 2
  Twitching | 1 | 1
  Headaches | 1 | 0
  Decreased appetite | 1 | 0
  Nausea | 0 | 1
  Hair loss | 1 | 0
  Fatigue | 1 | 0
  Flushed ears | 0 | 1
  Papules, rash | 1 | 0
  Double vision | 0 | 1
Statistical Analysis 1: Comparison: Placebo vs Naltrexone; Sleep disturbance; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 2: Comparison: Placebo vs Naltrexone; Unusual dreams; Test type: Superiority or Other; p = 0.45, Fisher Exact
Statistical Analysis 3: Comparison: Placebo vs Naltrexone; Twitching; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 4: Comparison: Placebo vs Naltrexone; Headaches; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 5: Comparison: Placebo vs Naltrexone; Decreased appetite; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 6: Comparison: Placebo vs Naltrexone; Nausea; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 7: Comparison: Placebo vs Naltrexone; Hair loss; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 8: Comparison: Placebo vs Naltrexone; Fatigue; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 9: Comparison: Placebo vs Naltrexone; Flushed ears; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 10: Comparison: Placebo vs Naltrexone; Papules, rash; Test type: Superiority or Other; p = 1.0, Fisher Exact
Statistical Analysis 11: Comparison: Placebo vs Naltrexone; Double vision; Test type: Superiority or Other; p = 1.0, Fisher Exact

ADVERSE EVENTS:
Groups:
- A: Placebo Control Group: Subjects will receive placebo for 8weeks
- B: Naltrexone, Active Drug Group: Naltrexone 0.1 mg/kg (not to exceed 4.5mg) once a day for 8 or 16 weeks
Arm/Group | A: Placebo Control Group | B: Naltrexone, Active Drug Group
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 5/6 | 4/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A: Placebo Control Group (N=6) | B: Naltrexone, Active Drug Group (N=12)
Sleep disturbance (Psychiatric disorders) | 2 | 2
Unusual dreams (Psychiatric disorders) | 0 | 2
Twitching (Nervous system disorders) | 1 | 1
Headaches (Nervous system disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Hair loss (Skin and subcutaneous tissue disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Flushed ears (Vascular disorders) | 0 | 1
Papules, rash (Skin and subcutaneous tissue disorders) | 1 | 0
Double vision (Eye disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
This was a pseudo-crossover trial where 6 subjects received placebo for 8 wks then were crossed over to active drug for 8 wks to increase the N treated with active drug. A smaller cohort of subjects on placebo were for safety & toxicity comparison.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No restrictions by the sponsor. The PI may disclose results after the manuscript has been published.